CLINICAL TRIAL: NCT06267222
Title: Trans-spinal Electrical Stimulation in Individuals With Spinocerebellar Ataxia: a Pragmatic Study
Brief Title: Trans-spinal Electrical Stimulation in Individuals With Spinocerebellar Ataxia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Laura Alice Santos de Oliveira (Other)
Collaborators: Federal Institute of Rio de Janeiro (Other)
Responsible Party: Sponsor-Investigator, Laura Alice Santos de Oliveira, Clinical Professor, Centro Universitário Augusto Motta
Organization: Centro Universitário Augusto Motta (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCATDCS23
Record Dates: First submitted 2023-10-11; First posted 2024-02-20 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: SCA; Postural Balance; Gait Ataxia
Keywords: NIBS; TRANS-SPINAL STIMULATION; CEREBELLAR ATAXIA
MeSH Terms: conditions — Gait Ataxia; Cerebellar Ataxia | interventions — Transcranial Direct Current Stimulation; Exercise Therapy

STUDY DESIGN:
Intervention Model Description: This is a pragmatic clinical trial that will be carried out using the CONSORT-Pragmatic Trials (Zwarenstein et al., 2008).
Masking Description: THE INVESTIGATOR NOT BE INFORMED ABOUT THE TREATMENT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- TRANS-SPINAL STIMULATION IN SCA (Experimental): The tDCS sessions will be conducted with an intensity of 2mA, utilizing the anodic electrode positioned over the cerebellar region and the cathodic electrode over the thoracic region of the spinal cord (approximately at vertebra T11). These sessions will be integrated into a gait and postural control training protocol, which will progressively increase in difficulty over 4 consecutive weeks on weekdays, excluding weekends. A total of 20 sessions will be administered, each lasting approximately 30 minutes. During each session, the electrodes will be placed, and participants will perform a single leg test on each side of the body. The exercise protocol will then be executed while the tDCS is applied, lasting for 20 minutes. Following the exercise, the single-leg test will be repeated, and the electrodes will be removed.
  Interventions: Device: TRANSCRANIAL DIRECT CURRENT STIMULATION + exercises

INTERVENTIONS:
Device: TRANSCRANIAL DIRECT CURRENT STIMULATION + exercises — Participants with SCA will receive trans-spinal tDCS and exercises. There will be no control group or sham stimulation. All participants will receive real tDCS stimulation
  Other Names: tDCS and exercises

SUMMARY:
The main goal of this pragmatic clinical trial is to investigate the effects of trans-spinal tDCS in individuals with spinocerebellar ataxia (SCA) over some parameters of gait and postural control in real-world conditions, reflecting daily clinical practice. The main questions it aims to answer are:

* If an extended number of tDCS sessions, beyond the typical 5 to 10 sessions described in scientific literature, applied concomitantly with exercises with progressive challenges, to yield positive outcomes over some parameters of gait and postural control in individuals with SCA and if there is retention of possible benefits one month later the end of this protocol.
* If there is specific characteristics (including balance, gait, mobility, severity of ataxia, DNA test characteristics and non-ataxic signs) in individuals with SCA that can predict their improvement in postural control and gait following the 20 tDCS sessions.

  * Participants will receive 20 tDCS sessions concomitantly with exercises for gait and postural control with progressive challenges.
  * Postural control and gait of the participants will be assessed in two big sessions before (#assessment 1) and after the 20 sessions (#assessment 5) and 3 small sessions after every 5 sessions (#assessments 2, 3 and 4). Also, as a follow-up, they will be assessed a month after the end of the intervention (#assessment 6).

DETAILED DESCRIPTION:
Spinocerebellar ataxias (SCA) comprise a group of progressive degenerative diseases, currently lacking pharmacological treatments. These conditions produce gait and balance disorders, ultimately necessitating the use of assistive devices, culminating in wheelchair dependency upon the loss of ambulatory function during the clinical progression of SCA. This significantly impacts the individual's independence and quality of life. Recent clinical trials have demonstrated that the application of transcranial direct current stimulation (tDCS) over the cerebellum and spinal cord (trans-spinal stimulation) has led to improvements in upper limb coordination, gait ataxia severity, motor scores (including balance), cognitive abilities, and quality of life in individuals with degenerative ataxias, including SCA. However, it is not yet known whether all patients with SCA demonstrate significant improvement with this intervention. Moreover, if there is no improvement, it remains unclear whether specific characteristics of individuals with SCA, such as balance, gait, mobility, ataxia severity, DNA test results, and non-ataxic signs, can be identified to predict their response to tDCS sessions. Additionally, tDCS studies in individuals with SCA typically involve 5 to 10 stimulation sessions without associating stimulation with exercises of progressive difficulty. One of the main benefits of using tDCS is the plastic modulation of the nervous system. Therefore, the lack of challenges concomitant with the use of tDCS limits its results. Aim: The main goal of this pragmatic clinical trial is to investigate the effects of trans-spinal tDCS in individuals with SCA over some parameters of gait and postural control in real-world conditions, reflecting daily clinical practice. The specific aims of this study are: (i) Determine whether particular characteristics of individuals with SCA (including balance, gait, mobility, severity of ataxia, DNA test characteristics and non-ataxic signs) can be identified to predict their improvement in balance and gait following tDCS sessions; (ii) to investigate if an extended number of tDCS sessions, beyond the typical 5 to 10 sessions described in scientific literature, applied concomitantly with exercises with progressive challenges, to yield positive outcomes over some parameters of gait and postural control in individuals with SCA; (iii) To investigate, through semi-structured interviews, the subjective experience of the participants regarding the use of trans-spinal tDCS, about changes in health and quality of life, as well as the expectations that were achieved or frustrated with the intervention used; (iv) To investigate if there is retention of benefits a month after the end of the intervention; (v) propose a specific test to detect postural control deficits during head and limb movement; and (vi) analyze whether the specific characteristics evaluated in individuals correlate with each other.

Methods: This is a pragmatic clinical trial that will be carried out using the CONSORT-Pragmatic Trials. The present study will be carried out at the Deolindo Couto Institute of Neurology, at the Federal University of Rio de Janeiro - UFRJ (Avenida Venceslau Brás, 95 - Botafogo, Rio de Janeiro - RJ). Individuals with spinocerebellar ataxia of any type, who are part of the records of public hospitals, doctors' offices, and physiotherapists, will be invited to participate in the study.

Initially, individuals will be interviewed to research the eligibility criteria, by filling out an anamnesis form, which will also contain questions about their demographic data. Those who are eligible and agree to participate must express their consent by signing an informed consent form.

Up to 45 patients with SCA of different types will undergo a non-invasive stimulation plus gait and postural control training. The total duration of sessions will last 30 minutes during which participants will simultaneously receive 20 min of trans-spinal tDCS and perform a gait training protocol with progressively greater difficulties, previously tested in patients with SCA. The trans-spinal tDCS will be applied at an intensity of 2mA, with the anodic electrode positioned over the cerebellar region and the cathodic electrode over the thoracic region of the spinal cord (approximately vertebra T11). The intervention will be applied over four consecutive weeks on weekdays except weekends, totaling 20 sessions.

All participants will receive real stimulation, so there will be no control group. Given that it may be difficult to recruit additional SCA individuals willing to participate in a control group or to find patients with similar characteristics who do not receive treatment during the study period, also due to the progressively debilitating condition of the participants (SCA) and given their socio-economic conditions that limit their transportation, it would be ethically questionable to deprive a group of patients of receiving a potentially beneficial treatment, especially when there is no established standard therapy or other effective treatment options available to them.

The equipment to be used for stimulation will be an NKL Stimulator. The continuous current offered will be supplied through a pair of 5x7 cm (35 cm2) electrodes wrapped in sponges moistened with saline solution. The anode electrode will be positioned over the cerebellar region. To do this, the inion region will be located. Using a measuring tape, the point 2cm above the inion will be identified and the electrode will be fixed to the scalp, using appropriate adjustable bands. The cathode electrode will be positioned over the spinal region, more precisely, at the level of T8. To precisely find this position, the thoracic spinous processes will be palpated, and the 11th process located. Using a measuring tape, identify the point located 2 cm below T11 and fix the electrode with adhesive tape at this point. The stimulation intensity will be 2mA.

Initially, participants will be evaluated (ASSESSMENT 1) through the application of the SARA scale; modified dynamic gait index (mDGI); The Berg Balance Scale; Timed up and go (TUG); Inventory of non-ataxic signs (INAS); The four-stage test; Ten-meter walk test with an accelerometer; and perform other three tasks using an accelerometer of a mobile phone: (i) 5 times sit-to-stand; (ii) Functional Reach Test; and (iii) a test consisted in move arms and head standing with foot together. Three physiotherapist experts in these evaluations who will not participate in the intervention sessions will conduct this part. Then, 20 successive tDCS sessions will be applied to the participants. Every 5 tDCS sessions, the mDGI and TUG assessment will be reassessed (ASSESSMENT 2, 3, and 4). At the end of the 20 sessions, all instruments will be reapplied except for INAS (ASSESSMENT 5). A month after the end of the intervention the individuals will be reassessed except for the tests using the accelerometer (ASSESSMENT 6).

Before and after each session, individuals will be evaluated using the one-leg stand test proposed in the miniBestest instrument. In this test, the individual must remain standing, with their eyes open and fixed on a point 1.6 to 3m away with their hands on their waist. The participant must remove a lower limb from the support, without assistance, flexing it backward and remaining there. The time spent in the position will be measured in seconds, from the moment the evaluator says "now" until the elevated foot touches the ground again, or the upper limbs move from the initial position. The test will be repeated twice for each lower limb. Both times will be noted, and the highest time will be considered.

At the end of 20 sessions, individuals who complete the intervention will be also interviewed with a semi-structurally questionary by a researcher who did not take part in the study. The method that will be used to analyze the interviews will be the framework approach, which consists of a deductive form of analysis that starts from pre-defined research objectives. The framework approach is a systematic method that allows for in-depth analysis, in which the researcher extracts codes from the interviewees' statements, forms categories, and finally acquires refined themes useful for describing the participants' ideas and perceptions. All interviews will be conducted face-to-face. The interviews will be recorded for future transcription, using a smartphone. Once the interviews have been transcribed, the content will be analyzed using ATLAS.ti® software, and, finally, the themes that most faithfully represent the concepts found in the interviews will be chosen.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 18 to 70, without distinction of gender or ethnicity;
2. Diagnosed with spinocerebellar ataxia, of any type, by a neurologist;
3. With mild to moderate ataxia severity;
4. Able to walk 2 meters even when using a walker, cane or crutch;
5. Score ≥21 (BERTOLUCCI et al., 1994) on the Mini-Mental State Examination (MMSE; FOLSTEINet al., 1975; ALMEIDA, 1998);
6. No other concomitant neurological changes.

Exclusion Criteria:

1. Illiterate;
2. Being subjected to any other experimental physiotherapeutic or medicinal intervention during the clinical trial;
3. Skin condition that may affect the electrode placement site
4. Musculoskeletal, neurological or cardiorespiratory disorders that prevent the tests from being carried out;
5. Epilepsy;
6. Pregnancy;
7. History of brain surgery;
8. History of seizures;
9. Metallic implants in the skull that interfere with neuromodulation;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Postural control | (i) Baseline, (ii) after 20 sessions and (iii) in follow up (one month).
  The Berg Balance Scale (BBS) measures functional balance and fall risk in 14 tasks. Each item is given a score of 0-4, with a total score between 0 and 56, being the higher the score, the better the individual's performance. The Berg scale also predicts the risk of falls. A score equal to or less than 45 points indicates a greater risk of falls.
  The four-stage test (4-stage) assesses static balance and measures an individual's ability to hold a series of four balance positions, each more challenging than the previous, for at least 10 seconds each.
Mobility | (ii) Baseline, (ii) at the end of sessions 5, 10, 15 and 20 (each session is 1 day) and (iii) in follow up (one month)
  Timed up and go (TUG) assesses mobility, balance, walking ability and the risk of falling. On the command "go", the patient gets up from the chair, walks 3 meters, turns around, returns to the chair, and sits down. The time is calculated in seconds. The longer the time taken, the greater the risk of falling
Gait performance | (ii) Baseline, (ii) at the end of sessions 5, 10, 15 and 20 (each session is 1 day) and (iii) in follow up (one month)
  Measured by the Modified Dynamic Gait Index (mDGI) which total score is from 0 (severe gait impairment) to 64 (no gait impairment) and a Ten-meter walk test with an accelerometer fixed at the sacrum to assess step and stride time, speed, and gait cadence.
Accelerometry | (i) Baseline and (ii) after 20 sessions.
  To perform three tasks using an accelerometer of a mobile phone fixed on the participant's waist: (i) 5 times sit-to-stand; (ii) Functional Reach Test; and (iii) a test consisted in move arms and head standing with foot together. The accelerometer will register how the body is moving and changing speed over time while performing tasks.

SECONDARY OUTCOMES:
The subjective experience of the participants regarding the protocol. | At the end of session 20 (each session is 1 day)
  Semi-structured interview regarding subjective experience of the participants relative to the study intervention
The presence of non ataxic signals (INAS) and the disease severity (SARA) | (i) Baseline and (ii) after 20 sessions.
  INAS is an inventary to detect the presence or absence of 16 non-ataxic signs and symptoms through a clinical physical examination. SARA is an instrument to evaluate the disease severity through eight tasks including gait, balance, speech and coordination that produce a total score of 0 (no signs of ataxia) and 40 (more severe ataxia).

CONTACTS AND LOCATIONS:
Overall Officials: LAURA OLIVEIRA, PT PHD, Study Director — Centro Universitário Augusto Motta; ANNA FONTES BAPTISTA, PT, Principal Investigator — Centro Universitário Augusto Motta; Eduardo S Moreira, PT, Study Chair — Centro Universitário Augusto Motta
Locations (1):
- Instituto de Neurologia Deolindo Couto, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Barretto TL, Bandeira ID, Jagersbacher JG, Barretto BL, de Oliveira E Torres AFS, Pena N, Miranda JGV, Lucena R. Transcranial direct current stimulation in the treatment of cerebellar ataxia: A two-phase, double-blind, auto-matched, pilot study. Clin Neurol Neurosurg. 2019 Jul;182:123-129. doi: 10.1016/j.clineuro.2019.05.009. Epub 2019 May 14. PMID 31121471
- [Background] Benussi A, Dell'Era V, Cotelli MS, Turla M, Casali C, Padovani A, Borroni B. Long term clinical and neurophysiological effects of cerebellar transcranial direct current stimulation in patients with neurodegenerative ataxia. Brain Stimul. 2017 Mar-Apr;10(2):242-250. doi: 10.1016/j.brs.2016.11.001. Epub 2016 Nov 3. PMID 27838276
- [Background] Benussi A, Dell'Era V, Cantoni V, Bonetta E, Grasso R, Manenti R, Cotelli M, Padovani A, Borroni B. Cerebello-spinal tDCS in ataxia: A randomized, double-blind, sham-controlled, crossover trial. Neurology. 2018 Sep 18;91(12):e1090-e1101. doi: 10.1212/WNL.0000000000006210. Epub 2018 Aug 22. PMID 30135258
- [Background] Benussi A, Batsikadze G, Franca C, Cury RG, Maas RPPWM. The Therapeutic Potential of Non-Invasive and Invasive Cerebellar Stimulation Techniques in Hereditary Ataxias. Cells. 2023 Apr 20;12(8):1193. doi: 10.3390/cells12081193. PMID 37190102
- [Background] Braga-Neto P, Godeiro-Junior C, Dutra LA, Pedroso JL, Barsottini OG. Translation and validation into Brazilian version of the Scale of the Assessment and Rating of Ataxia (SARA). Arq Neuropsiquiatr. 2010 Apr;68(2):228-30. doi: 10.1590/s0004-282x2010000200014. PMID 20464290
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Franchignoni F, Horak F, Godi M, Nardone A, Giordano A. Using psychometric techniques to improve the Balance Evaluation Systems Test: the mini-BESTest. J Rehabil Med. 2010 Apr;42(4):323-31. doi: 10.2340/16501977-0537. PMID 20461334
- [Background] Klockgether T, Mariotti C, Paulson HL. Spinocerebellar ataxia. Nat Rev Dis Primers. 2019 Apr 11;5(1):24. doi: 10.1038/s41572-019-0074-3. PMID 30975995
- [Background] Maas RPPWM, Toni I, Doorduin J, Klockgether T, Schutter DJLG, van de Warrenburg BPC. Cerebellar transcranial direct current stimulation in spinocerebellar ataxia type 3 (SCA3-tDCS): rationale and protocol of a randomized, double-blind, sham-controlled study. BMC Neurol. 2019 Jul 4;19(1):149. doi: 10.1186/s12883-019-1379-2. PMID 31272408
- [Background] Maia AC, Rodrigues-de-Paula F, Magalhaes LC, Teixeira RL. Cross-cultural adaptation and analysis of the psychometric properties of the Balance Evaluation Systems Test and MiniBESTest in the elderly and individuals with Parkinson's disease: application of the Rasch model. Braz J Phys Ther. 2013 May-Jun;17(3):195-217. doi: 10.1590/s1413-35552012005000085. PMID 23966138
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Matsuda PN, Taylor CS, Shumway-Cook A. Evidence for the validity of the modified dynamic gait index across diagnostic groups. Phys Ther. 2014 Jul;94(7):996-1004. doi: 10.2522/ptj.20130294. Epub 2014 Feb 20. PMID 24557650
- [Background] Orru G, Cesari V, Conversano C, Gemignani A. The clinical application of transcranial direct current stimulation in patients with cerebellar ataxia: a systematic review. Int J Neurosci. 2021 Jul;131(7):681-688. doi: 10.1080/00207454.2020.1750399. Epub 2020 Apr 7. PMID 32228395
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Schmitz-Hubsch T, Fimmers R, Rakowicz M, Rola R, Zdzienicka E, Fancellu R, Mariotti C, Linnemann C, Schols L, Timmann D, Filla A, Salvatore E, Infante J, Giunti P, Labrum R, Kremer B, van de Warrenburg BP, Baliko L, Melegh B, Depondt C, Schulz J, du Montcel ST, Klockgether T. Responsiveness of different rating instruments in spinocerebellar ataxia patients. Neurology. 2010 Feb 23;74(8):678-84. doi: 10.1212/WNL.0b013e3181d1a6c9. PMID 20177122
- [Background] Schmitz-Hubsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schols L, Szymanski S, van de Warrenburg BP, Durr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20. doi: 10.1212/01.wnl.0000219042.60538.92. PMID 16769946
- [Background] Woods AJ, Antal A, Bikson M, Boggio PS, Brunoni AR, Celnik P, Cohen LG, Fregni F, Herrmann CS, Kappenman ES, Knotkova H, Liebetanz D, Miniussi C, Miranda PC, Paulus W, Priori A, Reato D, Stagg C, Wenderoth N, Nitsche MA. A technical guide to tDCS, and related non-invasive brain stimulation tools. Clin Neurophysiol. 2016 Feb;127(2):1031-1048. doi: 10.1016/j.clinph.2015.11.012. Epub 2015 Nov 22. PMID 26652115
- [Background] Almeida OP. [Mini mental state examination and the diagnosis of dementia in Brazil]. Arq Neuropsiquiatr. 1998 Sep;56(3B):605-12. doi: 10.1590/s0004-282x1998000400014. Portuguese. PMID 9850757

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-10-11): https://cdn.clinicaltrials.gov/large-docs/22/NCT06267222/Prot_ICF_000.pdf